CLINICAL TRIAL: NCT06602037
Title: Development and Clinical Translation of immunoPET Imaging Probes for Pancreatic Cancer
Brief Title: ImmunoPET Imaging of Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2024-067-C
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Neoplasms Pancreatic
Keywords: Pancreatic cancer; ImmunoPET; Companion Diagnostics; Trop2; CLDN18.2（Claudin 18.2）; Gastric cancer; Solid tumors
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ImmunoPET imaging in patients with pancreatic cancers (Experimental): Enrolled pancreatic cancer patients (locally advanced or metastatic cancer) will undergo a Trop2/CLDN18.2-targeted immunoPET/CT scanning.
  Interventions: Diagnostic Test: [89Zr]Zr-DFO-SHR1920; Diagnostic Test: [18F]F-RESCA-3A12; Diagnostic Test: [68Ga]Ga-NOTA-3A12

INTERVENTIONS:
Diagnostic Test: [89Zr]Zr-DFO-SHR1920 — Enrolled pancreatic cancer patients will receive a single dose (1-3mCi) of [89Zr]Zr-DFO-SHR1920 (total 1-2mg antibody mass). Multiple immunoPET/CT imaging sessions will be performed on day 0, day 1(24 h), day 3 (72 h), day 5 (120 h) or day 7 (168 h).
  Other Names: [89Zr]Zr-SHR1920
Diagnostic Test: [18F]F-RESCA-3A12 — Enrolled pancreatic cancer patients will receive 0.05-0.1mCi/kg of [18F]F-RESCA-3A12. ImmunoPET/CT imaging will be acquired 1h after [18F]F-RESCA-3A12 injection.
  Other Names: [18F]F-3A12
Diagnostic Test: [68Ga]Ga-NOTA-3A12 — Enrolled pancreatic cancer patients will receive 0.05-0.1mCi/kg of [68Ga]Ga-NOTA-3A12. ImmunoPET/CT imaging will be acquired 1h after [68Ga]Ga-NOTA-3A12 injection.
  Other Names: [68Ga]Ga-3A12

SUMMARY:
Pancreatic cancer remains one of the most aggressive cancer types. Target-specific targeted therapy is an attractive therapeutic alternative for the treatment of patients with a wide range of cancers, including pancreatic cancer. Companion diagnostic technique is critical for the success of targeted therapies. SHR-A1921 is a TROP2-directed antibody-drug-conjugate (ADC) approved for several clinical trials for advanced solid tumors. SHR1920 is the humanized anti-Trop2 monoclonal antibody (hIgG1) of SHR-A1921. Radio-labeling SHR1920 with radionuclide Zirconium-89 (89Zr) enables non-invasive imaging and quantification of SHR-A1921 distribution in cancer patients. Performing a [89Zr]Zr-DFO-SHR1920 PET scan before treatment with SHR-A1921 can evaluate tracer uptake in the primary and metastatic tumor lesions and normal organ distribution. CLND18.2 is another potential therapeutic target for pancreatic cancer. Target-specific immunoPET imaging may help identify patients more likely to benefit from targeted therapy.

DETAILED DESCRIPTION:
Enrolled patients with pancreatic cancer will undergo whole-body [89Zr]Zr-DFO-SHR1920 immunoPET/CT scans at 0,1, 3, 5, or 7 days after tracer injection (1-3 mCi). Uptake of [89Zr]Zr-DFO-SHR1920 in tumor and normal organs/tissues will be scored visually and quantitatively. For immunoPET imaging with 18F or 68Ga-labeled 3A12 (a nanobody targeting CLDN18.2), immunoPET/CT scan will be performed 1h after tracer injection (0.05-0.1 mCi/kg).

Tumor uptake will be quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and accuracy will be calculated to evaluate the diagnostic efficacy. The correlation between lesion uptake and protein expression level determined by immunohistochemistry staining will be further analyzed. The exploration endpoint will be the imaging feasibility and preliminary diagnostic value of the above tracers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of pancreatic cancer or suspected pancreatic cancer by diagnostic imaging.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Known or suspected hypersensitivity to SHR1920, DFO/RESCA/NOTA, 89Zr/18F or 68Ga or any of the excipients.
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
SUV | 7 days
  Standardized uptake value (SUV) of [89Zr]Zr-DFO-SHR1920、[18F]F-RESCA-3A12 or [68Ga]Ga-NOTA-3A12 for each primary tumor of subject or suspected metastasis.
Biodistribution and radiation dosimetry of [89Zr]Zr-DFO-SHR1920 | 7 days
  Measurement of absorbed radiation doses to organs (Gy/MBq), tumour(s) and whole body (Sv/MBq).

SECONDARY OUTCOMES:
Sensitivity, Specificity, Positive predictive value (PPV), Negative predictive value (NPV) and accuracy | 30 days
  The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of [89Zr]Zr-DFO-SHR1920、[18F]F-RESCA-3A12 or [68Ga]Ga-NOTA-3A12 PET/CT will be calculated.
Trop2 expression and SUV | 30 days
  The Standardized uptake value (SUV) of [89Zr]Zr-DFO-SHR1920 will be calculated and the correlation between pathological results and tumor uptake of [89Zr]Zr-DFO-SHR1920 will be analyzed
CLDN18.2 expression and SUV | 30 days
  The Standardized uptake value (SUV) of [18F]F-RESCA-3A12 or [68Ga]Ga-NOTA-3A12 will calculated and the correlation between pathological results and tumor uptake of [18F]F-RESCA-3A12 or [68Ga]Ga-NOTA-3A12 will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Liu, PhD, Study Chair — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University; Weijun Wei, Ph.D. & M.D., Principal Investigator — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China